CLINICAL TRIAL: NCT02192840
Title: Regular DES Versus BiOSS Expert® Stent in Coronary Bifurcation Treatment - Randomized, Multicenter, Open-label, Controlled POLBOS I (POLish Bifurcation Optimal Stenting) Study
Brief Title: POLish Bifurcation Optimal Stenting Study
Acronym: POLBOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Collaborators: University National Heart Hospital (Other)
Responsible Party: Principal Investigator, Jacek Bil, MD, PhD, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.0
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Disease
Keywords: provisional T stenting; dedicated bifurcation stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon; Biosensing Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rDES Group (Active Comparator): Regular drug-eluting stent implantation, one of the following:
  Device: LucChopin (Balton, Poland) Device: Prolim (Balton, Poland) Device: Xience Pro (Abott Vascular) Device: Biomatrix (Biosensors) Device: Promus (Boston Scientific) Device: Cypher (Cordis) Device: Taxus (Boston Scientific) Device: Coroflex Please (BBraun) Device: Resolute Integrity (Medtronic)
  Interventions: Procedure: Coronary angioplasty with stent implantation
- BiOSS Group (Experimental): New dedicated bifurcation stent BiOSS Expert (Balton, Warsaw, Poland) implantation
  Interventions: Procedure: Coronary angioplasty with stent implantation

INTERVENTIONS:
Procedure: Coronary angioplasty with stent implantation — Coronary angioplasty in bifurcation lesion with drug-eluting stent implantation: BiOSS or regular DES (rDES)
  Other Names: Device: LucChopin (Balton, Poland); Device: Prolim (Balton, Poland); Device: Xience Pro (Abott Vascular); Device: Biomatrix (Biosensors); Device: Promus (Boston Scientific); Device: Cypher (Cordis); Device: Taxus (Boston Scientific); Device: Coroflex Please (BBraun); Device: Resolute Integrity (Medtronic)

SUMMARY:
Coronary bifurcation lesions pose therapeutic problems during percutaneous coronary interventions (PCI) and are associated with higher rates of periprocedural complications as well as higher rates of in-stent restenosis and stent thrombosis. Therefore the optimal approach to coronary bifurcations treatment is still a subject of debate, especially when the side branch is large, not easily accessible and narrowed by a long lesion. One of the proposed alternatives are dedicated bifurcation stents (DBS). However, there is large scarcity of randomized trials with DBS.

The aim of POLBOS I (POLish Bifurcation Optimal Stenting) study was to compare two intervention strategies for bifurcation treatment: provisional T-stenting (PTS) with any regular drug-eluting stent (rDES), the best treatment strategy at the moment, with stenting of bifurcation lesions with dedicated bifurcation paclitaxel-eluting stent BiOSS Expert® (Balton, PL).

ELIGIBILITY:
Inclusion Criteria:

* Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
* Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.

Exclusion Criteria:

* STEMI
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Subjects who refuse to give informed consent.
* Subjects with LVEF<30%
* Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
MACE | 12 months
  Cumulative rate of major adverse cardiovascular events (MACE) including cardiac death, myocardial infarction (MI) with or without ST-segment elevation and need for repeated revascularization of the target lesion (TLR).

SECONDARY OUTCOMES:
cardiac death | 12 months
all-cause death | 12 months
Target lesion revascularization | 12 months
Target vessel revascularization | 12 months
myocardial infarction | 12 months
late lumen loss | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Gil, MD, PhD, Principal Investigator — Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Locations (1):
- Department of Invasive Cardiology Central Clinical Hospital of the Ministry of Interior, Warsaw, Poland

REFERENCES:
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Vassilev D, Gil R. Clinical verification of a theory for predicting side branch stenosis after main vessel stenting in coronary bifurcation lesions. J Interv Cardiol. 2008 Dec;21(6):493-503. doi: 10.1111/j.1540-8183.2008.00400.x. Epub 2008 Oct 21. PMID 18973506
- [Background] Gil RJ, Vassilev D, Formuszewicz R, Rusicka-Piekarz T, Doganov A. The carina angle-new geometrical parameter associated with periprocedural side branch compromise and the long-term results in coronary bifurcation lesions with main vessel stenting only. J Interv Cardiol. 2009 Dec;22(6):E1-E10. doi: 10.1111/j.1540-8183.2009.00492.x. Epub 2009 Aug 20. PMID 19702678
- [Background] Vassilev D, Gil R, Kwan T, Nguyen T, Nanjundappa A, Doganov A. Extension distance mismatch--an unrecognized factor for suboptimal side branch ostial coverage in bifurcation lesion stenting. J Interv Cardiol. 2010 Aug;23(4):305-18. doi: 10.1111/j.1540-8183.2010.00574.x. Epub 2010 Jul 19. PMID 20642477
- [Background] Gil RJ, Vassilev D, Michalek A, Kern A, Formuszewicz R, Dobrzycki S, Wojcik J, Lesiak M, Kardaszewicz P, Lekston A. Dedicated paclitaxel-eluting bifurcation stent BiOSS(R) (bifurcation optimisation stent system): 12-month results from a prospective registry of consecutive all-comers population. EuroIntervention. 2012 Jul 20;8(3):316-24. doi: 10.4244/EIJV8I3A50. PMID 22829507
- [Derived] Gil RJ, Kern A, Formuszewicz R, Inigo Garcia LA, Dobrzycki S, Vassilev D, Bil J. 6-year results of BiOSS stents in coronary bifurcation treatment. Eur J Clin Invest. 2021 Aug;51(8):e13555. doi: 10.1111/eci.13555. Epub 2021 Mar 29. PMID 33782985